CLINICAL TRIAL: NCT01633814
Title: Influence of Hormone Replacement on Neural Cardiovascular Control in Postmenopausal Women
Brief Title: Hormone Replacement and Neural Cardiovascular Control in Postmenopausal Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution prior to completion of study. Data unavailable..
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1133919
Record Dates: First submitted 2012-06-25; First posted 2012-07-04 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-06

CONDITIONS: Menopause; Aging; Blood Pressure
Keywords: Physiological Processes; Exercise; Hormone replacement therapy
MeSH Terms: conditions — Motor Activity | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal estradiol (Experimental): Transdermal estradiol, delivery rate 100 µg day-1
  Interventions: Drug: Transdermal estradiol
- Placebo (Placebo Comparator): placebo patch.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Transdermal estradiol — transdermal estradiol, delivery rate 100 µg day-1
  Other Names: Elestrin
  Arms: Transdermal estradiol
Drug: Placebo — placebo patch.
  Arms: Placebo

SUMMARY:
Older women have an exaggerated increase in blood pressure during exercise. However, the reasons for this are unclear. It is important to investigate this phenomenon because a greater blood pressure response to exercise has been associated with an increased risk of stroke and mortality in otherwise healthy individuals. A unique aspect of aging in women is the profound change in hormone levels (i.e. estrogen and progesterone) associated with menopause. The influence of changes in estrogen and progesterone levels on the cardiovascular responses to exercise is poorly understood. However, it has been suggested that these hormones might change the responsiveness of the cardiovascular system. Possible mechanisms that could account for these changes are the arterial baroreflex and feedback from the exercising muscle (known as the exercise pressor reflex), both of which are known to powerfully modulate blood pressure during exercise. However, to date, few human studies have thoroughly examined the influence of changes in hormone levels on baroreflex function during exercise or the exercise pressor reflex in older women. As such, the purpose of this research project is to assess baroreflex function and the exercise pressor reflex in older women after transdermal estrogen and placebo.

DETAILED DESCRIPTION:
Study Design Older postmenopausal women will be randomized, in a double-blinded crossover design, to receive (i) transdermal estradiol, delivery rate 100 µg day-1 plus oral placebo, or (ii) placebo patch plus oral placebo. The experimental measurements and procedures below will be performed before and 4 weeks after each treatment.

Experimental measurements:

Blood Pressure- A blood pressure cuff will be wrapped around the right arm to obtain blood pressure via a standard automated auscultometric device (Welch-Allyn). In addition, beat-by-beat blood pressure will be obtained via finger photoplethysmography (Finapress blood pressure monitor).

Heart Rate- Standard limb lead electrodes will be used to obtain heart rate measurements.

Respiration- An elastic band will be placed around the subject's abdomen to measure rate and depth of breathing.

Blood Samples- A venous catheter will be placed in the subjects arm for blood samples. For screening purposes measurements of glucose, electrolytes, cholesterol and triglycerides will be made. In addition, progesterone, estrogen and testosterone, will be assessed to verify hormonal status.

Sympathetic Nerve Activity- A tiny microelectrode will be placed in the peroneal nerve of the leg, located just below the knee on the outer part of the leg. Alternatively, the median nerve located at the inside of the elbow will be used. At these points the nerves are closest to the surface of the skin. The course of the nerve will be determined by electrically stimulating through the skin with a pencil shaped electrode. When the nerve is stimulated, involuntary twitching and/or tingling sensations of the foot or hand will occur. The twitching or tingling will disappear when the stimulation is stopped. Once the nerve is found, two tiny, sterile, microelectrodes will be inserted through the skin. One is a reference electrode placed just above the nerve site (2 cm) and the other is the recording electrode. The recording electrode is advanced into the nerve. When the tip of the electrode enters the nerve, the subject may briefly notice either pressure or tingling sensations. At this point, minor adjustments in the position of the electrode will be made until an optimal nerve signal is obtained.

Limb Blood Flow Measurements- Blood flow to the arm or leg may also be measured by using duplex Doppler ultrasound to non-invasively measure mean arterial blood velocity and diameter. Femoral or brachial blood velocity can be obtained by placing a Doppler flow probe on the skin over the common femoral artery distal to the inguinal ligament or the brachial artery, respectively. Ultrasound imaging of femoral artery or brachial artery diameter will be performed at a site matching that at which velocity is measured. The following formula is used to calculate blood flow: blood flow = π * radius2 * velocity.

Urine samples will be collected to measure specific gravity and pH using test strips.

Experimental Procedures:

Neck Pressure and Neck Suction- A padded neck collar will be fitted around the anterior portion of the subject's neck for the application of brief 5-second periods of neck pressure and neck suction. This allows the application of positive or negative pressure to the carotid sinus baroreceptors which are located in this region. The positive pressure will transiently cause these receptors to detect a decrease in blood pressure and thus cause an acute increase in heart rate, and blood pressure. The negative pressure will transiently cause these receptors to detect an increase in blood pressure and thus cause an acute decrease in heart rate, and blood pressure. This procedure has been used extensively to non-invasively assess baroreflex function in healthy subjects aged between 18-80 years. Nevertheless, in subjects over 50 years of age Doppler imaging will be performed to screen for atherosclerotic plaques within the carotid vessels to rule out carotid artery disease and determine the feasibility of performing neck pressure and neck suction.

Handgrip Exercise and Post Exercise Ischemia- The subject will be asked to perform handgrip exercise for either two minutes or until they feel like they cannot maintain the exercise (i.e., fatigue). Five seconds before stopping the exercise, a cuff around the upper arm will be inflated to impede blood flow for 2 minutes. This traps the metabolites that were produced during the exercise in the area of the muscle, which maintains stimulation of skeletal muscle metaboreceptor afferents. Since these metaboreceptor afferents contribute to the rise in blood pressure during exercise, continued stimulation of these receptors maintains a blood pressure response.

ELIGIBILITY:
Inclusion Criteria:

* We plan to study female subjects of all ethnic backgrounds ranging in age from 18 to 80 years. Only healthy, normotensive individuals not taking medications will be included in this study.
* All postmenopausal women will be at least 4 years post menopause to avoid the potential for perimenopausal interference with study results

Exclusion Criteria:

* Active cardiopulmonary disease
* Hypertension
* Diabetes
* Chronic Obstructive Pulmonary Disease with concurrent daily use of inhalers.
* Known liver disease
* Peripheral neuropathy
* Chronic Kidney disease
* Pregnant women
* Any of the following contraindications to estrogen usage will cause exclusion:
* Personal or 1st degree relative (mother, sister, daughter) history of breast, ovarian, or uterine cancer
* Vaginal bleeding;
* Current thrombophlebitis or venous thromboembolic disorders including deep vein thrombosis or pulmonary embolus;
* Arterial thromboembolic disease such as stroke or myocardial infarction
* Migraine headaches
* Any previous intolerance to estrogen supplementation.
* Women who have smoked during the one-year period prior to enrollment.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Fadel, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total enrollment was 4 women. Study was terminated prematurely early due to poor enrollment and the fact that the PI was moving to another institution. No data was analyzed.
Groups:
- Transdermal Estradiol or Placebo: Transdermal estradiol, delivery rate 100 µg day-1 or placebo patch
  Transdermal estradiol: transdermal estradiol, delivery rate 100 µg day-1
Period: Overall Study
Arm/Group | Transdermal Estradiol or Placebo
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Total enrollment was 4 women. Study was terminated prematurely early due to poor enrollment and the fact that the PI was moving to another institution. No data was analyzed.
Arm/Group | Transdermal Estradiol or Placebo
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants] — Population: Total enrollment was 4 women. Study was terminated prematurely early due to poor enrollment and the fact that the PI was moving to another institution. No data was analyzed.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total enrollment was 4 women. Study was terminated prematurely early due to poor enrollment and the fact that the PI was moving to another institution. No data was analyzed.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotid Baroreflex Sensitivity (Bpm/mmHg)
Description: Carotid baroreflex sensitivity will be measured using the application of neck pressure and neck suction. Briefly, a variable neck pressure collar will be placed around the anterior two thirds of the neck to change carotid sinus transmural pressure.
Time Frame: Within one week prior to and then after one month of transdermal estrogen alone, transdermal estrogen plus progesterone, progesterone alone and placebo.
Population: Results are not available due to all members of the study having left the institution and not having made results available.
Arm/Group | Transdermal Estradiol or Placebo
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Exercise Pressor Reflex Responsiveness (Mean Blood Pressure Response (mmHg) and Muscle Sympathetic Nerve Activity Response (Burst Frequency) During Post Handgrip Ischemia.)
Description: To estimate exercise pressor reflex responsiveness changes in blood pressure and muscle sympathetic nerve activity from rest to during a period of post handgrip ischemia will be used.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Transdermal Estradiol or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Transdermal Estradiol or Placebo
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Total enrollment was 4 women. Study was terminated prematurely early due to poor enrollment and the fact that the PI was moving to another institution. No data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No